CLINICAL TRIAL: NCT05285930
Title: Effect of Bee Venom Phonophoresis on Healing of Chronic Lower Limb Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Mohamed othman, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/003573
Record Dates: First submitted 2022-02-28; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Ulcer, Leg
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Experimental): received phonophoresis with Bee Venom gel in form of a noncontact low-frequency pulsed ultrasound delivered through Bee Venom gel as a topical treatment at a distance of between 5 and 15 mm from the ulcer wound bed, and time was 10 minutes for each session in addition to conservative treatment of medical ulcer care.
  Interventions: Combination Product: Bee venom phonophoresis
- group B (Experimental): received phonophoresis with Bee Venom gel in form of a noncontact low-frequency pulsed ultrasound delivered through Bee Venom gel as a topical treatment at a distance of between 5 and 15 mm from the ulcer wound bed, and time was 10 minutes for each session in addition to conservative treatment of medical ulcer care.
  Interventions: Combination Product: Bee venom phonophoresis
- group C (Sham Comparator): received a noncontact low-frequency pulsed ultrasound delivered through only plain gel without BV gel at a distance of between 5 and 15 mm from the ulcer wound bed, and time was 10 minutes for each session in addition to conservative treatment of medical ulcer care.
  Interventions: Device: low intensity ultrasound

INTERVENTIONS:
Combination Product: Bee venom phonophoresis — phonophoresis with Bee Venom gel in form of a noncontact low-frequency pulsed ultrasound delivered through Bee Venom gel as a topical treatment at a distance of between 5 and 15 mm from the ulcer wound bed, and time was 10 minutes for each session in addition to conservative treatment of medical ulcer care. The performance of the ultrasound applicator was tested regularly before and after each patient exposure; each test included all relevant acoustic field parameters (pressure amplitude, frequency) and uniformity of the field distribution. This type of test of the acoustic output of the applicators was important to eliminate the possibility of any malfunctioning of the devices.
  Other Names: low intensity Ultrasound with bee venom gel
  Arms: group A; group B
Device: low intensity ultrasound — a noncontact low-frequency pulsed ultrasound delivered through plain gel only at a distance of between 5 and 15 mm from the ulcer wound bed, and time was 10 minutes for each session in addition to conservative treatment of medical ulcer care.
  Arms: group C

SUMMARY:
PURPOSE: to determine the impact of bee venom phonophoresis in accelerating ulcers healing.

BACKGROUND: Bee venom (BV) phonophoresis has been suggested as a noninvasive treatment for a number of inflammatory conditions and in healing of ulcers.

Ulceration due to vascular causes is often multifactorial and can be caused by both arterial and venous disease. Hypertension and atherosclerosis of the peripheral vessels lead to arterial disease associated with ischemic ulcers. Chronic venous insufficiency and the resulting venous hypertension cause venous ulcers.

There are lack in knowledge and information in published studies about the efficacy of bee venom phonophoresis as physical therapy modality in accelerating ulcers healing.

So, this study will be designed to provide a guideline about the efficacy of of bee venom phonophoresis in accelerating ulcers healing.

HYPOTHESES:

It will be hypothesized that:

It was hypothesized that Bee venom phonophoresis has no or limited effect in accelerating ulcers healing.

RESEARCH QUESTION: Does Bee venom phonophoresis an effect in accelerating ulcers healing?

DETAILED DESCRIPTION:
• A verbal explanation about the importance of this research procedure, main aims and conceptual approaches were explained to every participant. • Every participant was given his written informed consent for bee venom phonophoresis treatment • The procedures of this study were divided into two main parts: part one (measurement procedures) and part two (treatment procedures).

Bee venom allergy test: The participants had been tested for BV allergy; diluted BV, 0.05 ml, in normal saline (1 mg/ml) was injected intra-dermally into the forearm. If the tested lesion resulted in a wheal with a diameter of less than 10 mm and erythema with a diameter of less than 26.5 mm after 10 to 15 minutes, subjects were participated in this study.

1. Measurement procedure:

   A- Ulcer surface area Ulcer surface (UAS) would be calculated by placing a piece of sterilized transparency film over the ulcer and tracing the ulcer perimeter on the film with fine tipped transparency marker. A separate transparency was used for each Ulcer. The tracing is then placed over metric graph paper and the number of 1mm the tracing was counted (only full 1 millimeter squares inside the perimeter is counted and the area was converted to square centimeters).

   Ulcer area was measured before the beginning of the study and at the end of the first and second months of therapy and this process was repeated a minimum of three times for each measurement with the value obtained two or more times was reported.

   B-Ulcer volume measurement in cm3 (width x length x depth):
   * The patient would be positioned in a relaxed position with the ulcer directed upward.
   * The ulcer would be traced on transparent paper and placed over the metric graph paper to have the longest length and width.
   * A measuring tape would be directed into the deepest point of the ulcer to record the ulcer depth.
   * (width x length x depth)would be calculated to have the volume of the ulcer.

   B-Ulcer volume measurement in cm3 (width x length x depth):
   * The patient would be positioned in a relaxed position with the ulcer directed upward.
   * The ulcer would be traced on transparent paper and placed over the metric graph paper to have the longest length and width.
   * A measuring tape would be directed into the deepest point of the ulcer to record the ulcer depth.
   * (width x length x depth) would be calculated to have the volume of the ulcer
2. Treatment procedures:

Participants treated as outpatients, they were given information about the measurement and treatment procedures as well as about the bee venom phonophoresis before the beginning of the treatment, each participant history sheet was taken, they were asked to follow the surgeon and physical therapist instruction and asked to avoid heavy objects lifting as well as smoking.

Steps of the bee venom phonophoresis treatment procedures:

* Position of the participant: Put the participant in the most comfortable and relaxed position which is supine lying position then Remove any clothes above the abdomen to avoid restriction.
* Ultrasound device preparation: the plug of the ultrasound unit was inserted into the main current supply.
* Bee venom gel: the treatment approach (phonophoresis application for bee venom gel) had been prepared. Bee venom gel had been used for the study group and pure ultrasound gel had been used for the control group. Each participant received 0.6 mg up to maximum 1 mg BV gel each session • Phonophoresis application for bee venom gel (study group): A pulsed ultrasound (applicator 1.9 cm 2 ) had been applied around the incision site, the movement was over the incision margins with pulsed duty cycle 40% (4 ms on, 6 ms off), and Power density 0.5 W/cm2 and Time was 5 minutes each session. Treatment sessions were 3 sessions a week, for 3 consecutive weeks .
* Low intensity ultrasound with pure gel (control group): A low intensity pulsed ultrasound (applicator 1.9 cm 2 ) had been applied over the incision margins with pulsed duty cycle 20% (2 ms on, 8 ms off), and Power density 0.8 W/ cm 2 and Time was 5 minutes each session. Treatment sessions were 3 sessions a week, for 3 consecutive weeks 35 and medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients ranged in age from 40 to 60 years.
* They had not undertaken another physical therapy modality for ulcer healing
* non-smokers
* under their own prescribed medications, and controlled diet therapy as described by their physicians.
* All patients in the diabetic foot ulcer group (group B) were non-insulin dependent and had controlled blood glucose levels.

Exclusion Criteria:

* Patients with life-threatening disorders such as renal failure, myocardial infarction.
* any systemic diseases that may interfere with the study's objectives were excluded.
* patients with skin disease.
* any disease that can lead to ulcer rather than diabetes for the diabetic foot ulcer group only, as varicose veins, trauma, peripheral vascular diseases, and/or active malignancy.
* Ulcer with surface area of less than 2 cm2 or more than 8 cm2 would be excluded from the study.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
The ulcer surface area | changes from baseline, 6 weeks, 12 weeks of therapy.
  The ulcer surface area would be estimated by placing a piece of sterilized transparency film over the ulcer and using a fine-tipped transparency marker to trace the ulcer perimeter on the film. Each ulcer was treated with its own transparency. The trace was then placed on metric graph paper, and the count of 1mm squares within the perimeter was counted (only entire 1mm squares were counted, and the area was converted to square centimeters)
ulcer volume measurement | changes from baseline, 6 weeks, 12 weeks of therapy.
  The patient would be in a comfortable position, with the ulcer facing upward. To have the longest length and width, the ulcer would be traced on translucent paper and placed over the metric graph paper. A disposable measuring tape would be directed into the deepest point of the ulcer to record the ulcer depth. The volume of the ulcer would be calculated to have the width x length x depth ratio

CONTACTS AND LOCATIONS:
Overall Officials: eman othman, professor, Study Chair — Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in bee venom or ulcer . we will share the results of this study within 1 year following publication.
Supporting Information: SAP, ICF
Time Frame: 1 year after publication
Access Criteria: the criteria will be assessed by the publication of the trial in an international journals.

REFERENCES:
- [Derived] Othman EM, Hamada HA, Mohamed GI, Abdallah GA, Ahmed ZS, Al-Shenqiti AM, Kadry AM. Clinical and histopathological responses to bee venom phonophoresis in treating venous and diabetic ulcers: a single-blind randomized controlled trial. Front Med (Lausanne). 2023 Apr 20;10:1085544. doi: 10.3389/fmed.2023.1085544. eCollection 2023. PMID 37153087